CLINICAL TRIAL: NCT03376009
Title: A Study of Novel Biomarkers of Kidney Dysfunction in Patients Admitted for Liver Transplant Assessment.
Brief Title: A Study of Novel Biomarkers of Kidney Dysfunction at Liver Transplant
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC1
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Liver Transplantation; Liver Transplant; Complications; Kidney Dysfunction
Keywords: Biomarker
MeSH Terms: interventions — Blood Specimen Collection; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for serum and plasma Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant assessment patients: Adult patients admitted to the Scottish Liver Transplant Unit for liver transplant assessment, over a 6 month study period will be considered for recruitment.
  Interventions:
  Blood sample for serum and plasma biomarkers:
  Urine sample for biomarkers Cardiac bio-impedance (Cardioscreen Medis) Aortic pulse wave velocity (APWV) (TensioMed and SphygmoCor) Optical Coherence Tomography (Spectralis OCT) Arterial Spin Labelling Magnetic Resonance Imaging
  Interventions: Diagnostic Test: Blood sample for serum and plasma biomarkers:; Diagnostic Test: Urine sample for biomarkers; Diagnostic Test: Cardiac bio-impedance (Cardioscreen Medis); Diagnostic Test: Aortic pulse wave velocity (APWV) (TensioMed and SphygmoCor); Diagnostic Test: Optical Coherence Tomography (Spectralis OCT); Diagnostic Test: Arterial Spin Labelling Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Blood sample for serum and plasma biomarkers: — Serum/plasma biomarkers: Approximately 10ml (3 teaspoons) of blood will be extracted to measure pre-specified biomarkers of renal injury including kidney injury molecule-1 (KIM-1), cystatin C and neutrophil gelatinase-associated lipocalin (NGAL). Samples will then be stored to facilitate measurement of additional biomarkers in the future.
Diagnostic Test: Urine sample for biomarkers — Urinary biomarkers: A random urine sample will be obtained to measure urinary protein to creatinine ratio (uPCR), KIM-1 and liver-type fatty acid binding protein (L-FABP)
Diagnostic Test: Cardiac bio-impedance (Cardioscreen Medis) — Cardiac bio-impedance - a non-invasive assessment of cardiac output, cardiac index and systemic vascular resistance index using the bio-impedence technique (Cardioscreen 1000 Medis) Cardiac bio-impedance is performed by attaching sticky electrodes to the participant's neck and thorax. These electrodes pass a very low, constant and alternating current (1.5 mA, 86 kHz) across the thorax, which is imperceptible to the patient. This provides beat by beat data on cardiac output and haemodynamic measurements.
Diagnostic Test: Aortic pulse wave velocity (APWV) (TensioMed and SphygmoCor) — Aortic pulse wave velocity (APWV) a non-invasive measure of arterial function using oscillometric recordings to detail peripheral and central haemodynamics. This will be measured using two different techniques:
  TensioMed Arteriograph: After a rest period a blood pressure cuff inflates and deflates twice on the arm. This takes ~3 minutes and should cause only mild, temporary discomfort. The test will routinely be performed in duplicate to ensure accuracy of results.
  SphygmoCor: A pressure sensor is held over the radial pulse at the wrist to analyse the pulse wave. Then held over the carotid artery and/or femoral artery to assess the speed of the pulse wave through the body. The probe is similar to an ultrasound probe and should not cause any discomfort.
Diagnostic Test: Optical Coherence Tomography (Spectralis OCT) — OCT is a non-invasive imaging test which uses light waves to take cross sectional images of the back of the eye. Examination of the retinal and retinal nerve fibre layer thickness, macular volume, and choroidal thickness provides an assessment of generalised systemic microvascular injury. A strong correlation between choroidal thickness and renal dysfunction has previously been shown in patients with chronic kidney disease (Balmforth C et al, JCI Insight 2016).
  The participant is asked to sit in front of the OCT machine and rest their chin on a support to keep it motionless. The equipment will then scan the eye without touching it. Scanning takes about 5 - 10 minutes.
Diagnostic Test: Arterial Spin Labelling Magnetic Resonance Imaging — Magnetic resonance imaging using arterial spin labelling (ASL-MRI) This promising quantitative technique has the potential to identify dysregulated renal perfusion, stratify risk of AKI in pre-OLT patients, and to monitor alterations in renal haemodynamics in the post transplantation setting.
  * We aim to recruit 5 participants with 'normal' renal function (eGFR≥60ml/min/1.73m2) and a further 5 participants with 'abnormal' renal function (eGFR<60ml/min/1.73m2)
  * ASL-MRI will be performed in this subgroup during the week of OLT assessment and then repeated at 6-weeks post transplantation in those participants who undergo OLT during the study period.
  Other Names: ASL-MRI

SUMMARY:
Kidney dysfunction before and immediately after liver transplantation is common and leads to poorer outcomes, including prolonged need for post-operative intensive care, diminished graft survival, and greater risk of permanent kidney dysfunction and death. Blood creatinine level - the standard measure of kidney function - is suboptimal in people with advanced liver disease, overestimating kidney function by >20%. There is significant concern that liver transplant recipients are at higher risk of acute kidney injury (AKI) than we can currently predict. This study aims to identify superior tests (blood/urine or imaging) for kidney dysfunction, to enable improved treatment and patient outcomes.

This study aims to recruit 80-100 consecutive patients admitted to the Scottish Liver Transplant Unit (SLTU), Royal Infirmary of Edinburgh (RIE) for liver transplant assessment over a 6 month period. Permission will be sought to record the results of routine tests performed by the NHS during this assessment week. These tests include: electrocardiograph (ECG), Computed Tomography (CT) liver and abdomen, cardio-pulmonary exercise testing (CPEX), pulmonary function tests (PFTS), routine haematology and biochemistry blood tests, 24 hour urine collection and body composition analysis.

In addition, we will invite participants to attend the RIE clinical research facility (CRF) for a single visit (~2 hours) to perform extra research assessments. Blood and urine will be collected for biomarker analysis. Non-invasive assessment of cardiovascular function will be completed using cardiac bio-impedance and aortic pulse wave velocity. Examination of the blood vessels at the back of the eye will be performed using optical coherence tomography.

A subgroup of 10 participants will undergo magnetic resonance imaging (MRI) of the kidneys using arterial spin labelling to identify dysregulated renal perfusion. Patients who are transplanted during the study timeframe will be asked to re-attend the CRF for repeat assessments at 6 weeks post transplantation.

Funded by Scottish Liver Transplant Unit Endowment Fund

DETAILED DESCRIPTION:
Study population:

This prospective observational study will aim to recruit 80-100 consecutive patients admitted for liver transplant assessment to the Scottish Liver Transplant Unit in the Royal Infirmary of Edinburgh over a 6 month period.

Consent:

Potential participants will be identified by the clinical team involved in the patient's care. Thereafter, potentially suitable participants will be given information about the study both verbally (by a member of the research team) and in writing in the form of the patient information sheet. Potential patients will be given time (up to 24 hours) to consider their participation and discuss this with friends or family. If participants remain interested, written consent will be taken by the principal investigator or a suitably qualified and delegated member of the study site staff.

Study overview:

If the study entry criteria are met, and written consent is obtained the participant will be recruited to the study. Thereafter, permission will be sought to record the routine NHS administrative data (clinical, radiological and laboratory blood tests) that is collected as part of the routine NHS transplant assessment visit.

At a suitable time during the week long transplant assessment admission the participant will be transferred to theClinical Research Facility on the ground floor of the RIE for a 1-2 hour visit. During this study visit the following tests will be performed:

1. Blood tests:

   •Serum/plasma biomarkers: Approximately 10ml (3 teaspoons) of blood will be extracted to measure pre-specified biomarkers of renal injury including kidney injury molecule-1 (KIM-1), cystatin C and neutrophil gelatinase-associated lipocalin (NGAL). Samples will then be stored to facilitate measurement of additional biomarkers in the future. This point will be clear in the patient information sheet and consent form.
2. Urine tests:

   •Urinary biomarkers: A random urine sample will be obtained to measure urinary protein to creatinine ratio (uPCR), KIM-1 and liver-type fatty acid binding protein (L-FABP)
3. Imaging/monitors:

   * Cardiac bio-impedance - a non-invasive assessment of cardiac output, cardiac index and systemic vascular resistance index using the bio-impedence technique (Cardioscreen 1000 Medis) Cardiac bio-impedance is performed by attaching sticky electrodes to the participant's neck and thorax. These electrodes pass a very low, constant and alternating current (1.5 mA, 86 kHz) across the thorax, which is imperceptible to the patient. This provides beat by beat data on cardiac output and haemodynamic measurements.
   * Aortic pulse wave velocity (APWV) - a non-invasive measure of arterial function using oscillometric recordings at the brachial artery detailing both peripheral and central haemodynamics. This will be measured using two different technique (TensioMed Arteriograph and SphygmoCor)

   TensioMed Arteriograph: Aortic pulse wave velocity is performed by applying a blood pressure cuff to the participant's upper arm. After a rest period the test is started and the blood pressure cuff inflates and deflates twice. This process takes approximately three minutes and should cause only mild, temporary discomfort. The test will routinely be performed in duplicate to ensure accuracy of results.

   SphygmoCor: A pressure sensor is initially held over the radial pulse at the wrist to analyse the pulse wave. This sensor is then held over the carotid artery (side of the neck) and femoral artery (top of the leg) to assess the speed of the pulse wave through the body (pulse wave velocity). The probe is similar to an ultrasound probe and should not cause any discomfort to the patient.

   •Optical Coherence Tomography (OCT) (Spectralis OCT) -is a non-invasive imaging test which uses light waves to take cross sectional images of the back of the eye. Examination of the retinal and retinal nerve fibre layer thickness, macular volume, and choroidal thickness provides an assessment of generalised systemic microvascular injury. A strong correlation between choroidal thickness and renal dysfunction has previously been shown in patients with chronic kidney disease (Balmforth C et al, JCI Insight 2016).

   The participant is asked to sit in front of the OCT machine and rest their chin on a support to keep it motionless. The equipment will then scan the eye without touching it. Scanning takes about 5 - 10 minutes.

   In a subgroup of 10 patients:

   •Magnetic resonance imaging using arterial spin labelling (ASL-MRI) This promising quantitative technique has the potential to identify dysregulated renal perfusion and stratify risk of AKI in pre-OLT patients, and to monitor alterations in renal haemodynamics in the post transplantation setting.
   * We aim to recruit 5 participants with 'normal' renal function (eGFR≥60ml/min/1.73m2) and a further 5 participants with 'abnormal' renal function (eGFR<60ml/min/1.73m2)
   * In order to reduce the risk of selection bias we will approach consecutive patients to invite them to join this subgroup.
   * Weekly recruitment may be limited by scanner availability.
   * ASL-MRI will be performed in this subgroup during the week of OLT assessment and then repeated at 6-weeks post transplantation in those participants who undergo OLT during the study period.
   * Participants will be excluded if they have contra-indications to MRI.

   This test requires the participant to lie flat in the scanner for approximately 30 minutes. The participant will be able to talk to the professional performing the scan at all times, but they will not be allowed to move around whilst the scan is being performed. The participant will be asked to hold their breath for short periods of time (15-20 seconds) throughout the scan to allow image acquisition. Full details of this procedure will be given to the participant in the information leaflet. Those who are claustrophobic, who have an implantable device such as a pacemaker, and those who will find it prohibitively uncomfortable to lie in the scanner for approximately 30 minutes will be excluded from this subgroup.

   Participants who are transplanted during the timeframe of the study will be asked to attend the RIE CRF for a 1-2 hour follow-up visit at approximately 6-weeks post-transplantation (to coincide with their routine transplant clinic appointment).

   The following tests will be repeated:
   * Routine haematology and biochemistry tests
   * Biomarkers - urine/serum/plasma including uPCR
   * Cardiac bio-impedence
   * APWV
   * OCT
   * ASL-MRI - only if performed pre-transplant

   Morbidity data will be collected for all patients including need for renal replacement therapy (RRT) and change in renal function over time (ΔeGFR; change in estimated glomerular filtration rate).

   For those patients who receive a liver transplant during the 6 month study period; length of hospital stay, length of ITU admission, warm ischaemic time (time spent transplanting organ) and graft function will also be recorded.

   Mortality data will be obtained from Trak and transplant unit source data. Permission will be sought to obtain mortality data until 1-year post transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults over 18 years of age
* Able to provide written informed consent and able to understand and willing to comply with the requirements of the study
* Admission for assessment for liver transplantation

Exclusion Criteria:

* Patients who do not have capacity to consent
* Patients being assessed for liver transplantation because of acute liver failure
* Patients who are unwilling or unable to have an MRI scan will be excluded from the ASL-MRI study sub-group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who are admitted to the Royal Infirmary of Edinburgh (RIE) liver unit for liver transplant assessment over a 6-month period will be invited to join this study. They will be identified as potentially eligible by a member of their clinical care team, and thereafter will be introduced to a member of the research study team and given a participant information sheet. At present, approximately 4-5 patients are admitted for transplant assessment per week, therefore we anticipate that recruitment over a 6-month period would provide a potential of 80-100 participants.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Relationship between pre-transplant kidney function using novel biomarkers and post-transplant morbidity and mortality. | 6 months
  (KIM-1, NGAL, Cystatin C)

SECONDARY OUTCOMES:
Relationship between pre-transplant kidney perfusion using non-contrast ASL-MRI and pre-transplant renal dysfunction defined by eGFR | 7 days
  non-contrast Arterial spin labelling Magnetic Resonance Imaging (ASL-MRI)
Relationship between pre-transplant kidney perfusion using non-contrast ASL-MRI and post-transplant renal dysfunction defined by eGFR | 6 months
  non-contrast Arterial spin labelling Magnetic Resonance Imaging (ASL-MRI)
Relationship between pre-transplant cardiac bioimpedence and post-transplant renal dysfunction | 6 months
  Cardiac bioimpedence using cardioscreen medis
Relationship between pre-transplant APWV and post-transplant renal dysfunction | 6 months
  Aortic pulse wave velocity (APWV)
Relationship between pre-transplant plasma KIM-1 and post-transplant renal dysfunction | 6 months
  plasma KIM-1- biomarker of renal injury
Relationship between pre-transplant urinary protein to creatinine ratio and post-transplant renal dysfunction | 6 months
  urinary protein to creatinine ratio- urinary biomarker of renal injury
Relationship between retinal nerve fibre layer, choroidal thickness and pre-transplant renal function | 7 days
  Optical coherence tomography
Relationship between pre-transplant haemodynamic biomarkers and mortality at 1 year | 1 year
  Haemodynamic biomarkers as evidenced by cardiac bio-impedence, aortic pulse wave velocity +/- ASL-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Fallowfield, PhD, Principal Investigator — University of Edinburgh, NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised IPD that underlie results in a publication will be available only on direct request from another researcher